CLINICAL TRIAL: NCT01768208
Title: Metabolomic Variations in the Saxagliptin-Treated Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, the vice-president of Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CCEMD016
Record Dates: First submitted 2012-12-13; First posted 2013-01-15 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

ARMS (1):
- Saxagliptin (Experimental)
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin

SUMMARY:
This study is an open-label, cohort study to evaluate the potential mechanisms of Saxagliptin in the treatment of patients with type 2 diabetes (T2DM) using a comprehensive metabolomic method, in combination with fingerprint analysis and target analysis. It is a sub-study of STUDY: D168L00008.

ELIGIBILITY:
Inclusion Criteria:

* All the subject Inclusion Criteria should be referred to STUDY: D168L00008.

Briefly

1. Provision of informed consent prior to any study specific procedures
2. Diagnosed with type 2 diabetes
3. Men or women who are 18 years of age.
4. Patients should be drug naïve or treated with metformin alone on stable doses of for at least continues 8 weeks.
5. HbA1c are between 7.5% and 11.0%

Exclusion Criteria:

* All the subject Exclusion Criteria should be referred to STUDY: D168L00008.

Briefly

1. Pregnant or breastfeeding patients.
2. Insulin therapy within one year of enrolment(with the exception of insulin therapy during a hospitalization or use in gestational diabetes).
3. Previous treatment with any dipeptidyl peptidase-IV (DPP-IV) inhibitors or Glucagon-like peptide-1 (GLP-1) analogue.
4. History of administration of any antihyperglycemic therapy (other than metformin) during the 8 weeks prior to Visit 1(12 weeks for previous TZD).
5. Treatment with systemic glucocorticoids other than replacement therapy. Inhaled,local injected and topical use of glucocorticoids is allowed.
6. Treatment with strong cytochrome P450 inhibitors.
7. Gastrointestinal surgery that could impact the absorption of study drug.
8. Contraindications to therapy as outlined in the saxagliptin package insert.
9. Hypersensitivity to saxagliptin
10. Have a history of, or currently have, acute or chronic pancreatitis.
11. Type 1 diabetes, history of diabetic ketoacidosis or hyperosmolar non-ketonic coma.
12. Any condition where, in the opinion of the investigator, participation in this study may pose a significant risk to the patient or could render the patient unable to successfully complete the study.
13. Fasting plasma glucose >15mmol/l.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2012-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the changes in the metabolomic parameters before and after Saxagliptin treatment in type 2 diabetic patients. | 24 weeks
  The primary objective of the study is to compare the different metabolomic profiling at baseline (before treatment) and at the end of the study drug administration(24 weeks) using a Liquid Chromatography-Mass Spectrometry (LC-MS) analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China